CLINICAL TRIAL: NCT05856461
Title: Pulmonary Artery Denervation+ Atrial Fibrillation Ablation vs Atrial Fibrillation Ablation Only in Patients With Atrial Fibrillation and Group 2 of Pulmonary Hypertension
Brief Title: Pulmonary Artery Denervation in Patients With Atrial Fibrillation and Group 2 of Pulmonary Hypertension
Acronym: PADN+AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEN_02052023
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation; Pulmonary Hypertension
Keywords: Atrial fibrillation; Pulmonary Hypertension; Remote magnetic navigation; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation; Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: 2 parellel groups
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary vein isolation+sham pulmonary artery denervation (group 1) (Sham Comparator): In group 1, standard pulmonary vein isolation will be performed (with manual or remote robotic 3D navigation using radiofrequency energy) with sham pulmonary artery denervation procedure including 3D reconstruction of the pulmonary artery tree and creation of the false ablation point
  Interventions: Procedure: Pulmonary vein isolation; Procedure: Sham pulmonary artery denervation
- Pulmonary vein isolation+pulmonary artery denervation (group 2) (Active Comparator): In group 2, standard pulmonary vein isolation will be performed (with manual or remote robotic 3D navigation using radiofrequency energy) combined with pulmonary artery denervation procedure
  Interventions: Procedure: Pulmonary vein isolation; Procedure: Pulmonary artery denervation

INTERVENTIONS:
Procedure: Pulmonary vein isolation — Circumferential pulmonary vein isolation procedure using 3D navigation systems with entrance and exit block verification
Procedure: Sham pulmonary artery denervation — Sham pulmonary artery denervation procedure includes 3D reconstruction of the right ventricular outflow tract, main, left and right pulmonary arteries with creation of the false ablation points. No true ablation lesions will be performed in the pulmonary artery
  Arms: Pulmonary vein isolation+sham pulmonary artery denervation (group 1)
Procedure: Pulmonary artery denervation — Pulmonary artery denervation procedure includes 3D reconstruction of the right ventricular outflow tract, main, left and right pulmonary arteries and 3 circles of ablation lesions (bifurcation of the main pulmonary artery, left and right pulmonary arteries)
  Arms: Pulmonary vein isolation+pulmonary artery denervation (group 2)

SUMMARY:
The goal of the study is to compare efficacy and safety of the pulmonary artery denervation procedure combined with atrial fibrillation ablation versus atrial fibrillation ablation alone in patients with paroxysmal and persistent atrial fibrillation and group 2 of the pulmonary hypertension

ELIGIBILITY:
Inclusion Criteria:

* Mean pulmonary artery pressure > 25 mm Hg and pulmonary artery wedge pressure > 15 mm Hg by right heart catheterization
* Paroxysmal or persistent atrial fibrillation
* NYHA II-III
* BNP > 105 pg/ml
* Indications for catheter ablation of atrial fibrillation according guidelines
* LVEF > 50%

Exclusion Criteria:

* Group 1,3,4 of the pulmonary hypertension
* Left atrium diameter > 6 cm
* Planned open heart surgery procedure
* Previous heart valve surgery
* Severe aortic, pulmonary, tricuspid or mitral, valves regurgitation
* Thrombus in the left heart chambers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-12-29 (Estimated); Study Completion 2025-02-22 (Estimated)

PRIMARY OUTCOMES:
Freedom from Atrial Fibrillation/Atrial Flutter/Atrial Tachycardia | 12 months
  Freedom from Atrial Fibrillation/Atrial Flutter/Atrial Tachycardia 3 months after blanking period without antiarrhythmic drugs

SECONDARY OUTCOMES:
Perioperative complications | 30 days
  Perioperative complications, including Death, Stroke, TIA, myocardial infarction, cardiac tamponade, pulmonary vein stenosis, pulmonary vein stenosis, vascular complications
Clinical adverse events | 12 months
  Death, Stroke, TIA, myocardial infarction, cardiac arrest, bleedings
Number of hospitalizations | 12 months
  Hospitalizations due to atrial fibrillation of heart failure
Mean pulmonary artery pressure | 12 months
  Changes in mean pulmonary artery pressure between groups
Pulmonary vascular resistance | 12 months
  Changes in the pulmonary vascular resistance between groups
Pulmonary wedge pressure | 12 months
  Changes in the pulmonary wedge pressure between groups
Systolic pulmonary artery pressure | 12 months
  Changes in the systolic pulmonary artery pressure between groups
6-minutes walking distance | 12 months
  Changes in the 6-minutes walking distance between groups
Atrial fibrillation burden | 12 months
  Changes in the atrial fibrillation burden between groups
Brain natriuretic peptide | 12 months
  Changes in the brain natriuretic peptide between groups

CONTACTS AND LOCATIONS:
Overall Officials: Alexander B Romanov, MD, Principal Investigator — E. Meshalkin National Medical Research Center
Locations (1):
- E. Meshalkin National Medical Research Center, Novosibirsk, Russia